CLINICAL TRIAL: NCT00153140
Title: Polyethyleneglycol3350 vs Tegaserod in Treatment of Patients With Chronic Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 851-ZCC
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

INTERVENTIONS:
Drug: polyethyleneglycol3350

SUMMARY:
The purpose of this study is to compare the safety and efficacy of extended polyethyleneglycol3350 use to tegaserod in patients with chronic constipation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients at least 18 years of age
* Constipated according to ROME I criteria
* If female and of childbearing potential, patient must be surgically sterilized or using oral contraceptives, depot contraceptives, double- barrier method, intrauterine device, or testifies that she is monogamous with a vasectomized partner, or practices abstinence and will continue to do so during the duration of study
* Are otherwise in good health, as judged by a physical examination
* In the investigator's judgment, patient is mentally competent to sign an instrument of informed consent

Exclusion Criteria:

* Patients with heme positive stool at screening that is not associated with hemorrhoids or anal fissures.
* Patients with hypo- or hyperthyroidism as determined by medical history.
* Patients with severe renal impairment.
* Patients with moderate or severe hepatic impairment.
* Patients with known or suspected perforation or obstruction.
* History of gastric retention, inflammatory bowel disease, bowel resection, or colostomy.
* Patients with symptomatic gallbladder disease, suspected sphincter of Oddi dysfunction, or abdominal adhesions.
* Patients with a known history of organic cause for their constipation.
* Patients currently taking, or planning to take any of the following medications that are known to effect bowel habits:

  * Antidiarrheals
  * Antacids containing magnesium or aluminum salts
  * Anticholinergics
  * Antispasmodic agents
  * Erythromycin and other macrolides
  * Octreotide
  * Lotronex, Zofran, or other 5-HT3 antagonists
  * Zelnorm, or other 5-HT4 agonists
  * Opiods/narcotic analgesics
  * Prokinetics
  * Serotonin re-uptake inhibitors or tricyclic antidepressants
  * Calcium antagonists
* Patients who are breastfeeding, pregnant, or intend to become pregnant during the study.
* Female patients of childbearing potential who refuse a pregnancy test.
* Patients with a known allergy to tegaserod (or any of its excipients) or polyethyleneglycol.
* Patients who, in the opinion of the investigator, should not be included in the study for any reason, including inability to follow study procedures.
* Patients who, within the past 30 days have participated in an investigational clinical study.
* Patients that have undergone a colonoscopy within 30 days of screening
* Patients that are currently taking, or have previously been treated with polyethyleneglycol3350 or tegaserod.

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Enrollment: 239
Dates: Start 2004-07; Primary Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
A successful outcome is defined as no longer meeting the definition of constipation using ROME I criteria

SECONDARY OUTCOMES:
Analysis of individual ROME I criteria
Safety (adverse event review)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Herrera, MD, Principal Investigator — University of South Alabama
Locations (24):
- United States (24):
  - Mobile, Alabama
  - Glendale, Arizona
  - Anaheim, California
  - Sacramento, California
  - San Diego, California
  - Lake Worth, Florida
  - Largo, Florida
  - St. Petersburg, Florida
  - Laurel, Maryland
  - Brighton, Massachusetts
  - St Louis, Missouri
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Greer, South Carolina
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - San Angelo, Texas
  - Salt Lake City, Utah
  - Newport News, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia

REFERENCES:
- [Derived] Di Palma JA, Cleveland MV, McGowan J, Herrera JL. A randomized, multicenter comparison of polyethylene glycol laxative and tegaserod in treatment of patients with chronic constipation. Am J Gastroenterol. 2007 Sep;102(9):1964-71. doi: 10.1111/j.1572-0241.2007.01365.x. Epub 2007 Jun 15. PMID 17573794